CLINICAL TRIAL: NCT06171828
Title: Feasibility of Tele-education in Ultrasound Training: a Randomized, Controlled Pilot Study
Brief Title: Tele-education in Ultrasound Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2023-10-015-003
Record Dates: First submitted 2023-11-15; First posted 2023-12-15 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2023-11

CONDITIONS: Telemedicine; Ultrasonography; Education, Medical, Continuing
MeSH Terms: interventions — Smart Glasses

STUDY DESIGN:
Intervention Model Description: Interventional Clinical Trial, Parallel Assignment
Who Masked: Investigator
Masking Description: We plan to mask the identity of participant groups from the evaluators during the assessment process of the effectiveness of ultrasound education using tele-education. This blinding is intended to ensure the objectivity and integrity of the evaluation results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Traditional Training) (No Intervention): This arm of the study involves participants who will engage in a traditional learning process. After an initial pre-survey, they will start the ultrasound training phase. During this phase, participants will utilize pre-made educational videos for learning. Then participants will perform an ultrasound on an abdominal ultrasound phantom using a handout based on the pre-made video. When assistance is needed, participants will physically move to a different location to seek help from a supervisor. This face-to-face interaction allows for direct guidance and feedback. After completing the training sessions, participants will take a post-survey, which includes NASA-TLX, System Usability Scale (SUS), and a self-confidence assessment, to evaluate the training experience and measure the perceived workload, system usability, and confidence level changes due to the training.
- Experimental Group (Remote Training) (Experimental): In this arm, participants will undergo a remote learning process. Similar to the control group, they begin with a pre-survey followed by the training phase using the same educational videos. Participants view a handout on a head-mounted display(HMD) and perform an ultrasound on an abdominal ultrasound phantom. The key difference is that when they require assistance, they will use a HMD to communicate with a supervisor remotely. This allows the supervisor to provide guidance without being physically present, utilizing the HMD and potentially other remote communication tools for real-time interaction. The training phase is intended to mimic the in-person guidance as closely as possible through technological means. Following the training, the participants will also complete the same post-survey as the control group to assess the impact of remote training on their learning experience.
  Interventions: Device: Head-Mounted Display (HMD) to communicate with a supervisor remotely

INTERVENTIONS:
Device: Head-Mounted Display (HMD) to communicate with a supervisor remotely — Participants in the experimental group are oriented on using the education platform and communicating with the supervisor through an HMD for about 5 minutes. They then perform and save their ultrasound imaging. If they require assistance, they request help verbally through the HMD's communication system. The supervisor remotely observes and immediately assists upon request, utilizing the HMD and a 360-degree camera.
  Arms: Experimental Group (Remote Training)

SUMMARY:
The study aims to assess the impact of remote guidance in ultrasound training for medical professionals new to abdominal ultrasound. It involves 40 participants, divided into two groups of 20 each - a self-study group and a remote learning group. Participants include licensed doctors with no prior training in abdominal ultrasound, who are over 18 years old and have consented to participate.

DETAILED DESCRIPTION:
The study's design includes pre-surveys, random assignment, ultrasound training through educational videos, and distinct practice methods for each group - one with remote guidance and the other with traditional, in-person assistance. The effectiveness of training will be evaluated based on scores from evaluation forms, time taken for ultrasound imaging, frequency of requesting help, and surveys (NASA-Task Load Index, System Usability Scale, and a Self-confidence pre/post survey). Statistical analysis will be conducted using R software, employing tests such as the student t-test or Wilcoxon rank sum test.

This research is anticipated to provide valuable insights into the efficacy of remote guidance in ultrasound education, potentially influencing future medical training methodologies.

ELIGIBILITY:
Inclusion Criteria:

* Licensed doctor
* Participants who didn't receive prior training in abdominal ultrasound
* > 18 years old

Exclusion Criteria:

- Individuals who do not agree to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

PRIMARY OUTCOMES:
Ultrasound Skill Evaluation Scale | During the education session, approximately 30 minutes
  The composite scores from the evaluation forms will serve as the primary measure of effectiveness. These scores will be based on a standardized evaluation scale titled "Ultrasound Skill Evaluation Scale", which ranges from 0 to 90 points, where higher scores indicate better performance. Scores will be analyzed and compared using statistical tests such as the Student's t-test or the Wilcoxon rank-sum test to evaluate skill acquisition differences between groups.

SECONDARY OUTCOMES:
Ultrasound Imaging Duration | During the education session, approximately 30 minutes
  The time taken by participants from the moment they pick up the probe to begin the first image until they press the 'End Exam' button to save the final ultrasound image will be recorded and analyzed. This measure assesses efficiency and speed of learning, with comparison between groups using the Student's t-test or Wilcoxon rank-sum test.
Number of Assistance Requests | During the education session, approximately 30 minutes
  The frequency with which participants request help from the supervisor will also be tracked. This measure will help to understand the level of independence and confidence during the ultrasound procedure, as well as to determine if the time taken for the task is affected by these requests.

OTHER OUTCOMES:
NASA-Task Load Index (TLX) | After the training (Traditional and HMD), approximately 1hr
  The NASA Task Load Index (NASA-TLX) survey will be used to compare the perceived workload between participants seeking physical assistance and those receiving remote guidance through head-mounted displays (HMDs). Six aspects of workload will be assessed: mental demand, physical demand, temporal demand, performance, effort, and frustration. Scores range from 0 (lowest workload) to 100 (highest workload).
System Usability Scale (SUS) | After the training (Traditional and HMD), approximately 1hr
  Participants will complete the System Usability Scale (SUS) survey based on their experience with the abdominal ultrasound training. The SUS score measures system usability on a scale ranging from 0 to 100, with higher scores indicating better usability. The scores will be calculated according to the standard scoring system.
Confidence Assessment | After the training (Traditional and HMD), approximately 1hr
  Pre- and post-training surveys will assess participants' confidence in identifying abdominal organs using ultrasound. Confidence will be rated on a Likert scale from 1 (not confident at all) to 5 (extremely confident). Changes in self-perceived competence before and after training will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Meonghi Son, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
Not yet decided

REFERENCES:
- [Derived] Kim M, Son MH, Moon S, Cha WC, Jo IJ, Yoon H. A Mixed Reality-Based Telesupervised Ultrasound Education Platform on 5G Network Compared to Direct Supervision: Prospective Randomized Pilot Trial. JMIR Serious Games. 2025 Jan 16;13:e63448. doi: 10.2196/63448. PMID 39819654